CLINICAL TRIAL: NCT01569880
Title: Pre-flight Evaluation of Adult Patients With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CF-HAST-OUS
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-03

CONDITIONS: Cystic Fibrosis
Keywords: Blood gas response; Exercise; Gas exchange; Hypoxia altitude simulation test; Pulmonary function
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to investigate the relationship between hypoxemia achieved during Hypoxia Altitude Simulation test and sea level values of pulmonary function, arterial blood gases, pulse oximetry and cardiopulmonary exercise test variables. In addition, to study the effect of slow walk in a hypoxic environment, comparable to slow walking along the aisle.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis
* > 16 years
* Sputum test negative for Burkholderia cepacia and/or methicillin resistant Staphylococcus aureus

Exclusion Criteria:

* Ongoing infection

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with cystic fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Skrede, PhD MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Ullevål, Oslo, Norway

REFERENCES:
- [Derived] Edvardsen E, Akero A, Skjonsberg OH, Skrede B. Pre-flight evaluation of adult patients with cystic fibrosis: a cross-sectional study. BMC Res Notes. 2017 Feb 6;10(1):84. doi: 10.1186/s13104-017-2386-2. PMID 28166839